CLINICAL TRIAL: NCT00930358
Title: Tolerance and Acceptability of Colonoscopy Under Sedation by an Equimolar Mixture of Oxygen and Nitrous Oxide. Comparison With General Anesthesia in a Randomized, Multicentric Study.
Brief Title: Safety Study of Colonoscopy Under Sedation
Acronym: KALINAG
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was stopped due to low inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Cécile Kedzia, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060240
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Colonoscopy Procedure
Keywords: Sedation; Colonoscopy; General anesthesia
MeSH Terms: interventions — Meopa; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MEOPA (Experimental): MEOPA : equimolar nitrous oxide/oxygen mixture
  Interventions: Drug: MEOPA
- General anesthesia (Active Comparator): Gold standard
  Interventions: Drug: general anaesthesia

INTERVENTIONS:
Drug: MEOPA — anaesthetic gaz inhalation
  Other Names: anaesthetic gaz inhalation
  Arms: MEOPA
Drug: general anaesthesia — Anaesthetic intravenous route
  Other Names: Anaesthetic intravenous route
  Arms: General anesthesia

SUMMARY:
The aim of this study was to compare the analgesia provided by nitrous oxide/oxygen sedation or general anesthesia for colonoscopy

DETAILED DESCRIPTION:
The purpose of this protocol is to compare two methods of analgesia/sedation for colonoscopy. Sedation and analgesia induced by a 50% nitrous oxide/oxygen mixture could sufficient to allow the practice of colonoscopy instead of general anesthesia which is accompanied with certain risks and post procedure drowsiness.

ELIGIBILITY:
Inclusion Criteria:

1. Patient referred for colonoscopy with general anesthesia
2. Age above 18 et below 75 year
3. Patient who gave an informed consent

Exclusion Criteria:

1. Age below 18 ou above 75
2. Need for gastroscopy in the same procedure than colonoscopy
3. History of surgery wih resection more extended than half of the colon
4. Dementia with autonomy loss or psychiatric disorder non controlled by therapeutic
5. Severe congestive heart failure or evolutive heart ischemia
6. Recent cerebral stroke
7. Hemodynamic instability
8. Respiratory failure, severe chronic obstructive pulmonary (including asthma) or progressive pneumothorax
9. Hepatic failure (Child-Pugh score> 9)
10. Terminal renal failure 11 Hematopoietic disorders

12. Pathology with expected survival shorter than the duration of the study and cancer excepted basal cell carcinoma of the skin 13. Alcohol consumption higher than 100 gr per day 14. Pregnancy or breastfeeding at the inclusion period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who have well tolerated the colonoscopy as assessed by visual analogic scale (>75/100) | Immediately after the colonoscopy
The mean grade of patient anxiety before endoscopy | After the colonoscopy
  The mean grade of patient anxiety before endoscopy

SECONDARY OUTCOMES:
The mean tolerability of the colonoscopy between the group with sedation by nitrous oxide/oxygen mixture and the group with anesthesia | after the colonoscopy
The mean pain intensity during the procedure on a visual analogic scale | after the colonoscopy
The mean patient satisfaction on a visual analogic scale. | after the colonoscopy
The percentage of patients who agree to repeat the procedure in similar circumstances. | after the colonoscopy
The grade of difficulty of the colonoscopy evaluated by the endoscopist | After the colonoscopy
The mean duration of the endoscopy | After the colonoscopy
The percentage of caecum intubation | After the colonoscopy
The percentage of ileal intubation | After the colonoscopy
The opinion of the endoscopist on the tolerance of the colonoscopy | After the colonoscopy
The time to hospital discharge | After the issue of the colonoscopy
The Aldrete's score at the hospital discharge | After the colonoscopy
The number of patient who have refused the inclusion | After the issue of the colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Lamarque, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hotel Dieu Hospital, Paris, France

REFERENCES:
- [Background] Trojan J, Saunders BP, Woloshynowych M, Debinsky HS, Williams CB. Immediate recovery of psychomotor function after patient-administered nitrous oxide/oxygen inhalation for colonoscopy. Endoscopy. 1997 Jan;29(1):17-22. doi: 10.1055/s-2007-1004055. PMID 9083731